CLINICAL TRIAL: NCT03211845
Title: Pilot Study to Assess the Feasibility and Potential Impact of Nutritional Telemonitoring in Community Dwelling Elderly People Receiving Home Care
Brief Title: Feasibility of Nutritional Telemonitoring in Elderly Home Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: European Union (Other); Consorci Sanitari de Terrassa (Other); Viveris Technologies SA (Unknown); STMicroelectronics Grenoble 2 SAS (Unknown); Sirlan Technologies SAS (Unknown); Habitat Health Environment (Other); Universite Paris 13 (Unknown); Meditecnologia SA (Unknown); Cybermoor Ltd (Other); Telecom Sante (Unknown); Zorggroep Noordwest-Veluwe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL50423.081.14
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Undernutrition; Aging
Keywords: Ehealth; Older adults; Undernutrition; Feasibility study
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional telemonitoring (Experimental): Nutritional telemonitoring including self-measurements of body weight, nutritional status, appetite, diet quality and physical activity. Additionally, participants receive guidance on nutrition and physical activity by means of customized and general television messages and/or if necessary personal guidance by a nurse.
  Interventions: Other: Nutritional telemonitoring

INTERVENTIONS:
Other: Nutritional telemonitoring — Participants receive a weighing scale, pedometer and television channel in order to perform self-measurements and receive guidance on nutrition and physical activity. Nurses use a website in order to receive telemonitoring measurements and decide about proper follow-up. In case of risk of undernutrition, nurses provide personal advice to optimize nutritional status of the participant.

SUMMARY:
An optimal nutritional status is essential for healthy ageing. Telemonitoring might contribute to maintaining or improving nutritional status in elderly people.The objectives of this pilot study are to test the feasibility, acceptability and implementation fidelity of telemonitoring of nutritional parameters in community-dwelling older adults; to test the study procedures for effect evaluation; and to determine the likelihood of achieving desired impact on the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

Having a care referral for at least one of the following types of care:

* Domestic care
* Personal care
* Nursing care
* Individual or group support

Exclusion Criteria:

* Severe cognitive impairment (Mini Mental State Examination (MMSE) < 20)
* Receiving terminal care
* Expected length of receiving home care < three months
* Not having a television at home
* Clients with a visual impairment (not able to watch the television screen)
* Clients with a physical impairment in such a way, that they are not able to use the telemonitoring system
* Clients with nursing home care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-20 (Actual)

PRIMARY OUTCOMES:
Feasibility (qualitative outcome) | 12 weeks
  Qualitative outcome, measured using the process indicators acceptability, implementation, dose received, applicability. Data on these process indicators are collected using logbooks, semi-structured interviews, and questionnaires with items to be answered on a 5-point likert scale.

SECONDARY OUTCOMES:
Behavioural determinants | 12 weeks
  Measured by a self-developed questionnaire with statements concerning nutrition and physical activity to be answered on a 5-point likert scale.
Diet quality (DHD-index) | 12 weeks
  Measured by Dutch Healthy Diet index (DHD-index)
Nutritional status (MNA) | 12 weeks
  Measured by Mini Nutritional Assessment
Appetite (SNAQ) | 12 weeks
  Measured by Simplified Nutritional Appetite Questionnaire
Body weight (kg) | 12 weeks
  Measured by weighing scale of the brand A&D, type UC-411PBT-C
Physical functioning (SPPB) | 12 weeks
  Measured by Short Physical Performance Battery (SPPB)
Functional status (KATZ-15) | 12 weeks
  Measured by KATZ-15
Quality of life (SF-36) | 12 weeks
  Measured by Short-Form 36

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, Professor, Study Chair — Wageningen University and Research
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided